CLINICAL TRIAL: NCT05603637
Title: The Effect of Pulsed-field and Radiofrequency Ablation for Atrial Fibrillation on Platelet Activity, Coagulation and Inflammation
Brief Title: The Effect of Pulsed-field and Radiofrequency Ablation on Platelet, Coagulation and Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Pavel Osmancik, head of the department of arrhythmias, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PFA-RFA Thrombo
Record Dates: First submitted 2022-09-10; First posted 2022-11-02 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; radiofrequency ablation; pulsed-field ablation; platelet activity; coagulation
MeSH Terms: conditions — Atrial Fibrillation; Thrombosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation arm (Active Comparator): Patients will undergo pulmonary vein isolation by means of radiofrequency energy. The ablation will be done using SmartTouch ablation catheter (Biosense Webster, USA).
  Interventions: Procedure: Catheter ablation using SmartTouch radiofrequency ablation catheter
- Pulsed- field ablation arm (Experimental): Patients will undergo pulmonary vein isolation by means of pulsed-field ablation. The ablation will be done using Farawave ablation catheter (Boston Scientific, USA).
  Interventions: Procedure: Catheter ablation using Farawave pulsed-field ablation catheter

INTERVENTIONS:
Procedure: Catheter ablation using SmartTouch radiofrequency ablation catheter — Patients will undergo catheter ablation for atrial fibrillation, i.e. pulmonary vein isolation, using radiofrequency energy with SmatTouch ablation catheter (Biosense Webster, USA)
  Arms: Radiofrequency ablation arm
Procedure: Catheter ablation using Farawave pulsed-field ablation catheter — Patients will undergo catheter ablation for atrial fibrillation, i.e. pulmonary vein isolation, using pulsed-field energy with Farawave ablation catheter (Boston Scientific, USA)
  Arms: Pulsed- field ablation arm

SUMMARY:
The aim of the study is to compare platelet activation, activation of the coagulation and inflammation cascade during catheter ablation for atrial fibrillation using radiofrequency or pulsed-field energy. Patients with atrial fibrillation and standard indication for ablation according to the current guidelines will be randomized to ablation either using radiofrequency of pulsed-field energy. The endpoints will be parameters of platelet activation, activation of coagulation, and changes in inflammatory markers during ablation.

DETAILED DESCRIPTION:
Catheter ablation for atrial fibrillation (AF) , i.e. pulmonary vein isolation, is associated with the activation of platelets, coagulation cascade and inflammatory parameters. Thrombus in the left atrium could arise on sheaths or wires, but the highest risk presents the ablations itself. Radiofrequency ablation leads to immediate endocardial damage that presents strong pro-thrombotic milieu. To avoid thrombus formation on catheters in the left atrium, heparin with target activated clotting time (ACT) of 250-300 is given during the procedure.

Newly, pulsed - field ablation has been widely emerged. Since the pulsed-field energy presents substantially different kind of ablation energy, and the mechanism of action differs substantially (no thermal injury, no acute necrosis), also the effect on platelets, coagulation and inflammatory parameters could differ substantially.

The investigators therefore initiate a study comparing the effect of radiofrequency and pulsed-field ablation on parameters of platelet activation, coagulation and inflammation during catheter ablation.

Patients with AF indicated for catheter ablation according current guidelines will be randomized to radiofrequency or pulsed-field ablation. The procedure will be done using standard approach from one or both femoral veins under moderate analgesia. Using intracardiac echocardiography, and by means of SL1 sheath (Abbott, USA), transseptal puncture will be done. In patients in the radiofrequency arm, Lasso (circular mapping catheter) will be inserted in all four pulmonary veins, and using Smart Touch ablation catheter (Biosense Webster, USA), pulmonary vein isolation will be done with target ablation index of 400 on anterior and superior aspects of pulmonary veins and 350 of the posterior wall of the left atrium. In patients in the pulsed-field arm, SL1 sheath will be replaced by Faradrive sheath (Boston Scientific, USA), and pulmonary vein isolation will be done using Farawave catheter (Boston Scientific, USA).

Blood samples will be drawn at the beginning of the procedure from the right atrium (S1), after the transeptal puncture before the ablation from the left atrium (S2), after the ablation when all 4 pulmonary vein are isolated (S3), 24 hours after the procedure before patient discharge (S4), and 3 months after the procedure during follow-up.

Platelet activity will be determined using flow cytometry (membrane expression of P-selectin (CD62P) antigen, active part of the glycoprotein IIb/IIIa (PAC-1), CD 41/61 antigens). Changes in coagulation will be determined by measuring D-dimers and fibrin-monomers. Regarding the inflammatory parameters, plasma concentration of interleukin-6, and membrane activation antigens on leukocytes will be assessed using flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation - paroxysmal of persistent

Exclusion Criteria:

* pregnancy
* left atrium > 60 mm
* mechanical valve
* known prothrombotic state
* rheumatic heart disease
* severe valve disease (i.e. mitral insufficiency > 2, aortic stenosis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Membrane expression of CD62P | 3 months
  Platelet activity determined by activation marker
Membrane expression of PAC-1 | 3 months
  Platelet activity determined by activation marker
Concentration of D-dimers, fibrin-monomers,and voln Willebrand factor | 3 months
  Changes in the coagulation cascade
Concentration in interleukin-6 and membrane expression of leukocyte activation markers | 3 months
  CHanges in parameters of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be shared on demand
Supporting Information: Study Protocol
Time Frame: After study initiation

REFERENCES:
- [Derived] Osmancik P, Bacova B, Hozman M, Pistkova J, Kunstatova V, Sochorova V, Waldauf P, Hassouna S, Karch J, Vesela J, Poviser L, Znojilova L, Filipcova V, Benesova K, Herman D. Myocardial Damage, Inflammation, Coagulation, and Platelet Activity During Catheter Ablation Using Radiofrequency and Pulsed-Field Energy. JACC Clin Electrophysiol. 2024 Mar;10(3):463-474. doi: 10.1016/j.jacep.2023.11.001. Epub 2023 Nov 6. PMID 38085214